CLINICAL TRIAL: NCT04142112
Title: A Randomized, Blinded, Standard-Controlled, Study to Evaluate the Safety and Efficacy of Ohana In-Vitro Fertilization (IVF) Sperm Preparation Kit OHB035 on IVF
Brief Title: Randomized, Standard-Controlled, Study to Evaluate the Ohana IVF Sperm Preparation Kit, SPeRtility IVF Next Generation
Acronym: SPRING
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ohana BioSciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OHANA-IVF-001
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Infertility; Infertility, Male
MeSH Terms: conditions — Infertility; Infertility, Male | interventions — Reference Standards

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Ohana IVF Sperm Preparation Kit (Experimental): Samples in the Ohana IVF Sperm Preparation Kit group will undergo product-specific multistep processing in the lab prior to insemination.
  Interventions: Device: Ohana IVF Sperm Preparation Kit (OHB035)
- Standard IVF Preparation Kit (Active Comparator): Samples in the Standard IVF Sperm Preparation Kit group will undergo traditional processing in the lab prior to insemination.
  Interventions: Device: Standard IVF Preparation Kit (OHB037)

INTERVENTIONS:
Device: Ohana IVF Sperm Preparation Kit (OHB035) — The Ohana IVF Sperm Preparation Kit (OHB035) contains media for processing sperm through a series of timed steps prior to insemination with oocytes.
  Other Names: Ohana; OHB-035
  Arms: Ohana IVF Sperm Preparation Kit
Device: Standard IVF Preparation Kit (OHB037) — The Standard IVF Sperm Preparation Kit (OHB037) contains media for processing sperm per the traditional steps prior to insemination with oocytes.
  Other Names: Standard; OHB-037
  Arms: Standard IVF Preparation Kit

SUMMARY:
Multi-centered, randomized controlled study, evaluating the safety and efficacy of the Ohana IVF Sperm Preparation Kit vs. a standard IVF sperm preparation kit.

DETAILED DESCRIPTION:
This blinded, randomized, standard-controlled, paired study will be performed in approximately 83 healthy couples (pairs of male and female subjects), who are appropriate candidates for IVF in six fertility centers located in the United States (US).

The study will capture the selection of the best embryo for transfer and follow-up on pregnancy outcomes that result from the transfer of the selected embryo following the IVF procedure, and the results of safety assessments.

ELIGIBILITY:
Inclusion criteria: (Sample)

Female Inclusion Criteria:

1. Premenopausal, age 25-37 years at the time of providing informed consent, who is an appropriate candidate for IVF.
2. Infertility for ≥ 12 months with regular intercourse with current male partner (or >6 months if age >35).
3. Regular menses defined as 25 to 35-day cycles or an average of 10-13 spontaneous menstrual periods per year without exogenous hormones.
4. AMH between 1.8 - 4.9 ng/ml based on screening measurement at central laboratory.
5. AFC >14 within 3 months of screening visit.

Male Inclusion Criteria:

1. Willing and able to provide semen specimens at the Screening Visit and on the day of oocyte retrieval; (the specimen provided must be suitable for conventional IVF).
2. Provide a semen specimen with at least 4 million total motile sperm, following density gradient centrifugation and washing of the sample, at the Screening Visit.

Exclusion Criteria: (Sample)

Female Exclusion Criteria:

1. Recurrent pregnancy loss (defined as >2 clinical pregnancies without live birth).
2. Contraindications to being pregnant or to any of the IVF hormonal modulating medications to be used in this study.
3. History of severe ovarian hyperstimulation syndrome (OHSS) requiring medical or surgical intervention.
4. Clinically diagnosed polycystic ovarian syndrome (PCOS.)
5. Gynecologic history of: pelvic surgery (prior diagnostic or nonoperative laparoscopy, hysteroscopy or operative hysteroscopy are allowed.
6. Tobacco or nicotine use in the past 12 months.
7. History of substance abuse, including alcohol abuse.
8. Abnormal, undiagnosed, vaginal bleeding at the time of screening.

Male Exclusion Criteria:

1. History of: vasectomy or vasectomy reversal.
2. Inability and/or unwillingness to provide semen specimens.
3. Tobacco or nicotine use in the past 12 months.
4. History of substance abuse, including alcohol abuse.
5. Marijuana use in the past 12 months.

Ages: 25 Years to 37 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 83 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-11-26 (Estimated); Study Completion 2021-07-26 (Estimated)

PRIMARY OUTCOMES:
Blastocyst Evaluation | Three months following last patient treated.
  To compare the difference in the number of high-quality euploid blastocysts per mature oocyte in subjects undergoing split IVF insemination using sperm prepared with Ohana IVF sperm preparation kit OHB035 (OHANA) versus sperm prepared using a Standard IVF sperm preparation kit OHB037 (STANDARD)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Fertility Treatment Center, Tempe, Arizona
  - Women's Medical Research Group, LLC, Clearwater, Florida
  - Shady Grove Fertility, Rockville, Maryland
  - Boston IVF Fertility Clinic, Waltham, Massachusetts
  - Carolina Conceptions, P.A., Raleigh, North Carolina
  - Main Line Fertility Center, Bryn Mawr, Pennsylvania
  - Center for Assisted Reproduction, Bedford, Texas

IPD SHARING:
Plan to Share IPD: No
The data collected from this study will be pooled. The study size would not allow for statistical analysis on a site by site level.

REFERENCES:
- See also: Study sponsor webpage — http://ohanabio.com